CLINICAL TRIAL: NCT01845116
Title: Use of a Fish Oil-Based Intravenous Lipid Emulsion (Omegaven®) in the Treatment of Parenteral Nutrition (PN) Induced Liver Injury
Brief Title: Omegaven® in the Treatment of Parenteral Nutrition (PN) Induced Liver Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Omegaven 04-10-18B
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Results first posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-09

CONDITIONS: Total Parenteral Nutrition-induced Cholestasis
Keywords: PNALD; Cholestasis; Omegaven®; Short Bowel Syndrome
MeSH Terms: conditions — Cholestasis; Short Bowel Syndrome | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Single Omegaven® Intervention Arm
  Interventions: Drug: Omegaven®

INTERVENTIONS:
Drug: Omegaven® — 10% Omegaven® initiated at a starting dose of 0.5g/kg/day for two days and then advancing to the goal dose of 1g/kg/day, IV (in the vein) until the patient no longer requires parenteral nutrition or until participation in the study is terminated.
  Other Names: IV Fish Oil Based Lipid Emulsion

SUMMARY:
The purpose of this study is to determine whether the omega-3 fatty acid emulsion (Omegaven®), when used in place of the conventional soy-based fat emulsion (Intralipid), is effective in treating parenteral nutrition associated liver disease (PNALD) in children.

The study hypothesis is that Omegaven® can be safely provided to children who are dependent on parenteral nutrition and have PNALD, and can reverse or prevent progression of PNALD until the child can take adequate nutrition by mouth.

DETAILED DESCRIPTION:
Rationale for Omegaven® Treatment

Unlike conventional intravenous fat emulsions, Omegaven® is comprised solely of fish oils containing primarily omega-3 fatty acids. Animal studies have shown that IV lipid emulsions such as fish oil that are high in eicosapentaenic and docosahexaenoic acid reduce impairment of bile flow as seen in cholestasis caused by conventional fat emulsions(1,2). By administering Omegaven® in place of conventional phytosterol/soybean fat emulsions, the cholestasis may be reversed and patients will be able to be maintained on adequate PN until they are able to ingest adequate nutrition enterally.

References

1. Chen W. Effects of fat emulsions with different fatty acid composition on plasma and hepatic lipids in rats receiving total parenteral nutrition. Clinical Nutrition 1996;15:24.
2. Yeh S. Effects of fish oil and safflower oil emulsions on diet-induced hepatic steatosis in rats receiving total parenteral nutrition. Clinical Nutrition 1996;15:80.

ELIGIBILITY:
Inclusion Criteria:

* Children 0-18 years of age
* Patients will be PN-dependent and expected to continue PN for at least 30 days
* Patients considered eligible for study participation must have PN-associated liver diseases . Other causes of liver disease (i.e., biliary atresia, galactosemia, alpha-1 antitrypsin deficiency) will be excluded. A liver biopsy is not necessary for treatment
* Direct bilirubin > 2.0 mg/dl
* Signed patient informed consent
* Signed patient assent where applicable.

Exclusion Criteria:

* Pregnancy
* Other causes of chronic liver disease (cystic fibrosis, biliary atresia, alpha-1 antitrypsin deficiency)
* Signs of advanced liver disease including cirrhosis on biopsy, varices, ascites
* The patient is allergic to eggs/shellfish
* The patient has a severe hemorrhagic disorder
* The patient is enrolled in any other clinical trial involving an investigational agent (unless approved by the designated physicians on the multidisciplinary team)
* The parent or guardian or child unwilling to provide consent or assent.

Ages: 4 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A. Caicedo, MD, Principal Investigator — Levine Children's Hospital at Carolinas HealthCare System
Locations (1):
- Levine Children's Hospital at Carolinas HealthCare System, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Upon study completion

REFERENCES:
- [Background] Puder M, Valim C, Meisel JA, Le HD, de Meijer VE, Robinson EM, Zhou J, Duggan C, Gura KM. Parenteral fish oil improves outcomes in patients with parenteral nutrition-associated liver injury. Ann Surg. 2009 Sep;250(3):395-402. doi: 10.1097/SLA.0b013e3181b36657. PMID 19661785
- [Background] Gura KM, Lee S, Valim C, Zhou J, Kim S, Modi BP, Arsenault DA, Strijbosch RA, Lopes S, Duggan C, Puder M. Safety and efficacy of a fish-oil-based fat emulsion in the treatment of parenteral nutrition-associated liver disease. Pediatrics. 2008 Mar;121(3):e678-86. doi: 10.1542/peds.2007-2248. PMID 18310188
- [Background] Gura KM, Duggan CP, Collier SB, Jennings RW, Folkman J, Bistrian BR, Puder M. Reversal of parenteral nutrition-associated liver disease in two infants with short bowel syndrome using parenteral fish oil: implications for future management. Pediatrics. 2006 Jul;118(1):e197-201. doi: 10.1542/peds.2005-2662. PMID 16818533

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Normalization of Direct Bilirubin
Description: Normalization of direct bilirubin is defined as less than 0.4mg/dL by 9 months.
  This relates to the efficacy of parenteral administration of fish oil derived fat emulsion (Omegaven®) to reverse established parenteral nutrition associated liver disease.
Time Frame: Month 9
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 11
participants | 11

2. Secondary Outcome: Number of Participants With Normal Essential Fatty Acid (EFA) Profiles.
Description: EFA is defined at a triene tetraene ratio of greater than 0.2 (so normal is > 0.2). Collected monthly from month 1-9.
Time Frame: Months 1 through 9
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 11
Participants | 10

3. Secondary Outcome: Number of Participants With Triglyceride Levels > 400 mg/dL
Description: Number of participants with triglyceride levels > 400 mg/dL
Time Frame: baseline data and then weekly and monthly evaluations, for an average of 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 11
Participants | 0

4. Secondary Outcome: Number of Participants With Unexpected Bleeding or Coagulopathies
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 11
Participants | 0

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=11)
Essential fatty acid deficiency (Metabolism and nutrition disorders) | 1 (1) — One patient had a mild essential fatty acid deficiency and went off Omegaven but had already achieved reversal of cholestasis.

LIMITATIONS AND CAVEATS:
The last patient enrolled in the study was on 11/8/2016. Due to decreased enrollment permission was granted by the Atrium Health IRB to officially close the study to new enrollees on May 31, 2019. The last patient enrolled is now 5 years removed from enrollment date.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2010-07-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT01845116/Prot_000.pdf
  • Informed Consent Form (2010-07-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT01845116/ICF_001.pdf